CLINICAL TRIAL: NCT03924778
Title: Modifying Diet and the Gut Microbiota to Reduce Obesity and Health Disparities
Brief Title: Modifying Diet to Improve Gut Microbiome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003207
Record Dates: First submitted 2019-03-25; First posted 2019-04-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH diet (Experimental): calorie-restricted DASH diet (25% fat; 57% carbohydrate; 18% protein; 34 g fiber
  Interventions: Behavioral: DASH diet
- standard American diet (Active Comparator): calorie-restricted standard American diet (35% fat; 51% carbohydrate; %15 protein; 14 g fiber
  Interventions: Behavioral: standard American diet

INTERVENTIONS:
Behavioral: DASH diet — brief description
  Arms: DASH diet
Behavioral: standard American diet — describe
  Arms: standard American diet

SUMMARY:
The investigators will conduct a 2-arm randomized controlled pilot, feasibility feeding study in which 28 participants will be randomized to receive either a calorie-restricted Dietary Approaches to Stop Hypertension (DASH) diet or a calorie-restricted standard American diet provided by the study for 4 weeks. Participants will be non-Hispanic black or white, generally healthy females (14 black, 14 white). The investigators will collect fecal samples at multiple time points before, during, and after the dietary intervention to analyze for changes in the gut microbiota and functional-level metabolic products. This work will be led by an interdisciplinary team including expertise in bio-behavioral science, microbiology, nutrition science, bioinformatics, and biostatistics all with cross-cutting expertise in health disparities, prevention research, nutrition, the gut microbiota, inflammation and other biomarkers. The rationale for the proposed research is that once the interactions between race, diet, and the gut microbiota are more fully understood, targeted diet modifications may provide new and innovative approaches for the prevention and treatment of obesity and obesity-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* female
* non-Hispanic, black or white
* age 19-65 years
* BMI >= 30 kg/m^2
* able to visit Bionutrition Unit daily

Exclusion Criteria:

* gastrointestinal (GI) conditions i.e., irritable bowel, diverticulitis, peptic ulcers, Crohn's, GI cancers, and adenatomous polyps
* antibiotic or probiotic use in the previous 90 days
* tobacco use
* heavy alcohol consumption
* major medical conditions (e.g., renal disease, diabetes, cancer)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean Weight Change of Participants | Baseline to day 28
  Weight change as measured by a scale in kilograms at multiple time points will be calculated and averaged.
Mean Weight Change of Participants | Day 28 to Day 42
  Weight change as measured by a scale in kilograms at multiple time points will be calculated and averaged.
Mean Weight Change of Participants | Baseline to day 42
  Weight change as measured by a scale in kilograms at multiple time points will be calculated and averaged.
Diet-specific changes in secondary bile acid | Baseline to day 28
  The investigators will calculate changes in cholic acid in milligrams.
Diet-specific changes in secondary bile acid | day 28 to day 42
  The investigators will calculate changes in cholic acid in milligrams.
Diet-specific changes in secondary bile acid | baseline to day 42
  The investigators will calculate changes in cholic acid in milligrams.
Diet-specific changes in inflammatory marker | baseline to day 28
  The investigators will calculate changes in c-reactive protein in mg/L.
Diet-specific changes in inflammatory marker | day 28 to day 42
  The investigators will calculate changes in c-reactive protein in mg/L.
Diet-specific changes in inflammatory marker | baseline to day 42
  The investigators will calculate changes in c-reactive protein in mg/L.
Diet-specific changes in short chain fatty acids | baseline to day 28
  The investigators will calculate changes in acetic acid in mmol/L
Diet-specific changes in short chain fatty acids | day 28 to day 42
  The investigators will calculate changes in acetic acid in mmol/L
Diet-specific changes in short chain fatty acids | baseline to day 42
  The investigators will calculate changes in acetic acid in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany L Carson, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffit Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No